CLINICAL TRIAL: NCT06998394
Title: A Single-Arm, Phase II Clinical Trail of Cadonilimab Combined With Chemoradiotherapy in Oligometastatic Stage IVB Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangbo Wan (Other)
Responsible Party: Sponsor-Investigator, Xiangbo Wan, doctor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-1629-003
Record Dates: First submitted 2025-03-05; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer Stage IV
Keywords: Cadonilimab; Cervical Cancer; Oligometastasis; Individualized Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AK104 (Experimental)
  Interventions: Drug: AK104 - Chemotherapy

INTERVENTIONS:
Drug: AK104 - Chemotherapy — AK104 (10mg/kg, q3w) + cisplatin weekly or every 3 weeks + radiotherapy (pelvic external beam radiotherapy + brachytherapy) until disease progression, intolerable toxicity, or the investigator judgment that the participant can no longer benefit, participant withdrawal of consent, or completion of 2 years of AK104 treatment.

SUMMARY:
Cervical cancer is one of the most malignant reproductive system tumors that threaten women's health, characterized by distinct HPV-driven carcinogenesis and immunosuppressive tumor microenvironment. According to statistics from the World Health Organization (WHO) and the GLOBOCAN database, there were approximately 604,127 new cases of cervical cancer worldwide in 2022, with about 341,831 deaths, accounting for 6.5% of all female cancer-related deaths. While HPV vaccines can effectively reduce the incidence of cervical cancer, which has demonstrated 90% efficacy in preventing HPV16/18-associated malignancies, the global incidence and mortality rates of cervical cancer have not shown a significant downward trend. Cervical cancer also has a high recurrence rate, with approximately 30% of intermediate and advanced cervical cancer cases recurring within 5 years, and the 5-year survival rate for high-risk patients after recurrence is less than 20%. It is evident that cervical cancer remains a serious threat to women's health. Current research has confirmed that more than 90% of cervical cancer cases are associated with persistent infection with high-risk HPV viruses. HPV-positive status is positively correlated with increased PD-L1 expression, and PD-L1 expression in cervical cancer tissues is closely related to the proliferation and activation of CD8+ T cells. Preclinical models demonstrate that dual checkpoint blockade PD-1/CTLA-4 inhibition synergistically enhances CD8+ T cell activation and tumor regression in HPV+ cervical cancer xenografts. Therefore, cervical cancer patients are likely to benefit from immunotherapy. Based on the unmet treatment needs of cervical cancer and its high immune response, immunotherapy for cervical cancer has become a focus of attention in the field of gynecological oncology in recent years. The pharmacokinetics, and immunogenicity characteristics of this regimen, provide an effective treatment option to further improve the survival of advanced cervical cancer patients.

Based on the above research background, this study targets stage IVB cervical cancer with oligometastasis. In addition to systemic chemotherapy combined with individualized radiotherapy, cadonilimab, one bispecific antibody for PD-1/CTLA-4, is added to explore the preliminary anti-tumor activity, safety, pharmacokinetics, and immunogenicity characteristics of this regimen, providing an effective treatment option to further improve the survival of advanced cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Capacity Participants must be able to understand and voluntarily sign a written informed consent form. The informed consent form must be duly signed before any study-specific procedures are performed.
2. Demographic Parameters Female participants aged ≥ 18 years on the day of signing the informed consent form.
3. Functional Status Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Prognostic Threshold Expected survival ≥ 6 months.
5. Diagnostic Confirmation Histologically or cytologically confirmed cervical cancer.
6. Lesion Quantification At least one measurable tumor lesion according to RECIST v1.1 criteria.
7. Biomarker Accessibility All participants must be willing to provide tumor tissue samples before enrollment.
8. Organ Functional Reserve

   Screening laboratory values meeting the following thresholds (performed within 7 days prior to enrollment):
   1. Hematopoietic: ANC ≥1.5×10⁹/L; Platelets ≥100×10⁹/L; Hemoglobin ≥9 g/dL.
   2. Hepatic: Total bilirubin ≤1.5×ULN; AST/ALT ≤2.5×ULN.
   3. Renal: Serum creatinine ≤1.5×ULN OR calculated CrCl ≥60 mL/min (Cockcroft-Gault).
9. Reproductive Safety

Women of childbearing potential (WOCBP) must:

1. Demonstrate negative serum β-hCG pregnancy test within 72 hours prior to treatment initiation.
2. Utilize dual contraceptive methods (e.g., oral contraceptives + barrier device) from screening through ≥120 days post-final dose and ≥180 days post-chemoradiation.
3. Abst requiresinence declaration medical confirmation non of-reproductive status.

Exclusion Criteria:

1. Histopathological Exclusions

   1. Participants with other histological types of cervical cancer, such as neuroendocrine carcinoma, small cell carcinoma, sarcoma, etc.
   2. Mixed epithelial-mesenchymal tumors with >50% non-squamous component.
2. Orange State Exclusions

   1. History of total hysterectomy (removal of the uterine body and cervix). Subtotal hysterectomy or cornual resection with preservation of the cervix is allowed.
   2. Anatomical abnormalities or tumor geometry-related contraindications that prevent the use of brachytherapy.
   3. Clinically significant bilateral hydronephrosis that cannot be relieved by nephrostomy or ureteral stenting, as judged by the investigator.
3. Oncological History Other active malignancies within 2 years before enrollment, except for locally curable cancers that have been cured, such as squamous cell carcinoma of the skin, basal cell carcinoma of the skin, superficial bladder cancer, and breast carcinoma in situ.
4. Therapeutic Exposure

   1. Previous treatment with immune checkpoint inhibitors or any tumor immunotherapy targeting immune co-stimulatory factors.
   2. Use of systemic corticosteroids (> 10 mg/day prednisone or equivalent doses of corticosteroids) or other immunomodulatory drugs within 2 weeks before enrollment.
   3. Use of live vaccines within 4 weeks before enrollment.
   4. Major surgery within 4 weeks before enrollment (as determined by the investigator), open biopsy, or significant trauma; or planned major surgery during the study. Systemic pelvic/para-aortic lymphadenectomy for diagnostic purposes is allowed.
5. Concomitant Disease Exposure

   1. Active infections requiring systemic treatment, or active autoimmune diseases, except for vitiligo, alopecia, psoriasis, or eczema not requiring systemic treatment; hypothyroidism caused by autoimmune thyroiditis requiring only stable hormone replacement therapy; type 1 diabetes requiring only stable insulin replacement therapy.
   2. Known primary or secondary immunodeficiency, including positive human immunodeficiency virus (HIV) antibody test.
   3. Active or documented history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), active diverticulitis.
6. Past Medical History Exposure

   1. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
   2. Known history of interstitial lung disease or non-infectious pneumonia.
   3. Known history of severe hypersensitivity to monoclonal antibodies.
7. Cardiovascular Diseases Exposure

   1. Myocardial infarction, unstable angina, pulmonary embolism, aortic dissection, deep vein thrombosis, or any arterial thromboembolic event within 6 months before enrollment.
   2. Heart failure with New York Heart Association (NYHA) class ≥ II.
   3. Severe arrhythmias requiring long-term drug intervention; asymptomatic atrial fibrillation with stable ventricular rate is allowed.
   4. Cerebrovascular events (CVA) within 6 months before enrollment.
   5. Left ventricular ejection fraction (LVEF) < 50%.
   6. History of myocarditis or cardiomyopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-3-year progression-free survival | From enrollment to 3 years after the end of treatment

SECONDARY OUTCOMES:
Objective response rate | at least 12 weeks
Disease control rate | at least 12 weeks
Overall survival | From date of randomization until the date of death，assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- 1 Jianshe East Road, Erqi District, Zhengzhou City, Henan Province, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes